CLINICAL TRIAL: NCT06243653
Title: The Role of Coronary Microvascular Dysfunction in Improving Left Ventricular Systolic Function Using Registry for Evaluation of Factors associatEd With Heart Failure With Reduced Ejection Fraction Caused by Non-ischemic Etiology (REFERENCE).
Brief Title: Relationship Between Coronary Microvascular Dysfunction and Improvement of Left Ventricular Systolic Function in Patients With Heart Failure With Reduced Ejection Fraction Caused by Non-ischemic Etiology
Acronym: HFrEF-CMD
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: HFrEF-CMD
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Microvascular Angina; Non-ischemic Cardiomyopathy
Keywords: coronary microvascular dysfunction; non-ischemic cardiomyopathy
MeSH Terms: conditions — Heart Failure; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFrEF: Patients with heart failure with reduced ejection fraction (HFrEF) without significant coronary artery disease (non-ischemic cardiomyopathy)
  Interventions: Diagnostic Test: CMD test

INTERVENTIONS:
Diagnostic Test: CMD test — Measured CFR and IMR
  Other Names: Coronary microvascular dysfunction

SUMMARY:
This study aims to evaluate the incidence of coronary microvascular dysfunction (CMD) and its prognostic implication for the improvement of left ventricular function in patients who have been diagnosed with heart failure with reduced ejection fraction (HFrEF) caused by non-ischemic etiology.

DETAILED DESCRIPTION:
HF is a clinical syndrome characterized by dyspnea or exertional limitation due to impairment of ventricular filling or ejection of blood or both. HFrEF occurs when the left ventricular ejection fraction (LVEF) is 40% or less and is accompanied by progressive left ventricular dilatation and adverse cardiac remodeling. Among them, a substantial portion of patients had non-ischemic etiology.4 The CMD, defined by impaired coronary flow reserve (CFR), is commonly observed in patients with cardiomyopathies caused by non-ischemic etiology and is well-known to be associated with poor prognosis independently of the degree of left ventricular functional abnormality. However, the presence of CMD can be more specifically evaluated by invasive physiologic assessment using both CFR and the index of microcirculatory resistance (IMR) than by non-invasive methods (doppler echocardiography, positron emission tomography, or cardiac magnetic resonance imaging [MRI]) measuring CFR alone. Considering that CMD, defined by depressed CFR with elevated IMR, reflects the impaired myocardial flow and microvascular damages, there was a possibility that it may be a predictor of irreversible myocardial damages in HFrEF patients with non-ischemic etiology. Nevertheless, there has been limited data regarding the association between the improvement of LV function and CMD for patients with HFrEF caused by non-ischemic etiology after guideline-directed medical treatment (GDMT). Therefore, the investigators sought to evaluate the incidence of CMD and its prognostic implication for the improvement of left ventricular function after GDMT in patients who have been diagnosed with HFrEF caused by non-ischemic etiology.

ELIGIBILITY:
Inclusion Criteria:

* a) Subject must be at least 19 years of age. b) Subject with symptoms or signs of HF (NYHA ≥2 dyspnea) and reduced ejection fraction (LVEF ≤ 40%) c) Subject who clinically need coronary angiography d) Subject who can voluntarily sign informed consent form

Exclusion Criteria:

* a) Subject with significant coronary artery stenosis on coronary angiography (diameter stenosis ≥90% or 50-90% with fractional flow reserve [FFR] ≤0.80) b) Subject scheduled for cardiac replacement therapy (heart transplantation or left ventricular assisted device [LVAD] implantation) c) HF due to restrictive cardiomyopathy, active myocarditis, or constrictive pericarditis d) Significant valvular heart disease requiring surgery e) Subject who have non-cardiac co-morbid conditions with life expectancy <1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with reduced ejection fraction (HFrEF) without significant coronary artery disease (non-ischemic cardiomyopathy)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of HFiEF* at 12 months | 1-year follow-up
  HFiEF was defined as LVEF >40% measured by echocardiography at 12 months.1

SECONDARY OUTCOMES:
Correlation between CMD and left ventricular end diastolic pressure | 1 year
Correlation between CMD and delta LVEF from baseline to 12 months | 1 year
Correlation between CMD and E/e' | 1 year
Correlation between CMD and delta LV systolic dimension from baseline to 12 months | 1 year
Correlation between CMD and delta LV diastolic dimension from baseline to 12 months | 1-year follow-up
Correlation between CMD and late gadolinium enhancement measured by cardiac MRI | 1 year
Correlation between CMD and pulmonary artery wedge pressure | 1 year
Correlation between CMD and mean pulmonary artery pressure | 1 year
Correlation between CMD and pulmonary artery pulsatility index (PAPi) | 1 year
Correlation between CMD and cardiac output/cardiac index | 1 year
Correlation between CMD and delta NT-proBNP from baseline to 12 months follow-up | 1-year follow-up
Proportion of CMD according to etiology | 1 year
Rates of All-cause death | 1-year follow-up
Rates of Cardiac death | 1-year follow-up
Rates of Readmission due to HF | 1-year follow-up
Rates of Readmission | 1-year follow-up
Rates of Implantation of implantable cardioverter defibrillator | 1-year follow-up
Rates of Cardiac replacement therapy (heart transplantation or LVAD) | 1-year follow-up
Changes of quality of life for HF (Kansas City Cardiomyopathy Questionnaire [KCCQ]) | 1-year follow-up
Total medical cost | 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hong Choi, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea